CLINICAL TRIAL: NCT00527306
Title: Prevention of Recurrent Aphthous Stomatitis Using Vitamins
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Rajesh Lalla, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-022-1; DF 04-005 (Other Grant/Funding Number: Donaghue Medical Research Foundation)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Aphthous Stomatitis
Keywords: aphthous stomatitis; canker sores; multivitamins; vitamin deficiency
MeSH Terms: conditions — Stomatitis, Aphthous; Avitaminosis | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I - Multivitamin (Experimental): The multivitamin will contain 100% of the US reference daily intakes (recommended daily amounts) of vitamins A, B1, B2, B3, B5, B6, B9, B12, C, D, and E. It also contains several inactive ingredients including sodium bisulfite and gelatin.
  Interventions: Dietary Supplement: multivitamin
- II - Inactive Medication (Placebo Comparator): The placebo will be a gelatin capsule filled with lactose.
  Interventions: Dietary Supplement: multivitamin

INTERVENTIONS:
Dietary Supplement: multivitamin — Subject will be asked to take a multivitamin capsule or a placebo (inactive pill) once a day for one year. There will be an equal chance of getting the multivitamin or the placebo.

SUMMARY:
The purpose of this research study is to find out if taking a multivitamin daily can affect the number of canker sores that people get and how long they last. Previous studies have shown that people who get canker sores are more likely to be deficient in one or more vitamins. It has also been found that correction of such vitamin deficiencies reduces the number and duration of canker sores. However, it is not known if taking a multivitamin daily will reduce the number and duration of canker sores.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to provide written informed consent for the study
* Patients with a history of at least three episodes of minor recurrent aphthous stomatitis (RAS) within the past one year

Exclusion Criteria:

* Patients with a history of other forms of RAS (major, herpetiform)
* Patients who will be using any other vitamins/supplements during the study or those who have used any vitamins/supplements on a regular basis during the 90 days immediately preceding enrollment onto the study (regular use is defined as continuous daily use for at least a two week period)
* Patients who are under the age of 18
* Women who are pregnant or nursing or those who plan to become pregnant
* Patients with a history of gout, kidney stones or iron overload disease
* Patients who currently smoke tobacco products
* Patients who are former smokers who have quit smoking within the past 30 days
* Patients with sulfite allergy
* Patients with a history of any systemic condition associated with oral ulceration. These include: Behcet's syndrome, Sweet's syndrome, Celiac disease, Crohn's disease, ulcerative colitis, HIV infection/AIDS, cyclic neutropenia and PFAPA syndrome (periodic fever, aphthous stomatitis, pharyngitis and cervical adenitis)
* Patients on medications commonly associated with causing oral ulceration. These include nicorandil, methotrexate and chemotherapeutic agents used for cancer.
* Patients using oral topical anti-inflammatory agents during the course of the study
* Patients who plan to use any products specifically for management of RAS lesions
* Patients who are routinely using agents that could have an impact on duration of RAS lesions (e.g., antibacterial mouthrinses)
* Patients receiving any other investigational agent during the course of ths study
* Patients with any other condition that might preclude participation in the study in the opinion of the study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Annual number and average duration of minor recurrent aphthous stomatitis (canker sores) episodes | one year

SECONDARY OUTCOMES:
Pain due to recurrent aphthous stomatitis (canker sores); impact of recurrent aphthous stomatitis on ability to consume a normal diet | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh V. Lalla, DDS,PhD,CCRP, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Result] Lalla RV, Choquette LE, Feinn RS, Zawistowski H, Latortue MC, Kelly ET, Baccaglini L. Multivitamin therapy for recurrent aphthous stomatitis: a randomized, double-masked, placebo-controlled trial. J Am Dent Assoc. 2012 Apr;143(4):370-6. doi: 10.14219/jada.archive.2012.0179. PMID 22467697
- [Result] Huling LB, Baccaglini L, Choquette L, Feinn RS, Lalla RV. Effect of stressful life events on the onset and duration of recurrent aphthous stomatitis. J Oral Pathol Med. 2012 Feb;41(2):149-52. doi: 10.1111/j.1600-0714.2011.01102.x. Epub 2011 Nov 12. PMID 22077475
- [Result] Kozlak ST, Walsh SJ, Lalla RV. Reduced dietary intake of vitamin B12 and folate in patients with recurrent aphthous stomatitis. J Oral Pathol Med. 2010 May;39(5):420-3. doi: 10.1111/j.1600-0714.2009.00867.x. Epub 2010 Feb 7. PMID 20141576
- See also: Publication describing results of this study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3880249/
- See also: Publication describing results of this study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3323121/
- See also: Publication describing results of this study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3323114/